CLINICAL TRIAL: NCT06170515
Title: Performance Evaluation of Blood Glucose Meters and HbA1c Point-of-care Devices
Brief Title: BGM and HbA1c POC Device Evaluation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NC002
Record Dates: First submitted 2023-10-27; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Arm 1: Evaluation of BGM's (listed below)
  * CareSens N-Eco (i-Sens)
  * CareSens N-Premier (i-Sens)
  * CodeFree (SD Biosensor)
  * GlucoNavii GDH (SD Biosensor) Comparator BGMs: Ascensia Contour Next One and Nova Statstrip Xpress (BG); using strip lots meeting CLSI POCT12 acceptance criteria as validated at an experienced laboratory using traceable analysers
  Arm 2: HbA1c evaluation (listed below)
  * Affinion (Abbott)
  * HbA1c 501 (HemoCue)
  * A1Care (iSens)
  * DCA Vantage (Siemens)
  Reference: NGSP-certified HbA1c laboratory method, validated with ERL reference samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BGM Evaluation (Other)
  Interventions: Diagnostic Test: CareSens N-Eco (i-Sens), • CareSens N-Premier (i-Sens), CodeFree (SD Biosensor), GlucoNavii GDH (SD Biosensor)
- HbA1c evaluation (Other)
  Interventions: Diagnostic Test: Affinion (Abbott), HbA1c 501 (HemoCue), A1Care (iSens), DCA Vantage (Siemens)

INTERVENTIONS:
Diagnostic Test: CareSens N-Eco (i-Sens), • CareSens N-Premier (i-Sens), CodeFree (SD Biosensor), GlucoNavii GDH (SD Biosensor) — BGM Test
  Arms: BGM Evaluation
Diagnostic Test: Affinion (Abbott), HbA1c 501 (HemoCue), A1Care (iSens), DCA Vantage (Siemens) — HbA1c Test
  Arms: HbA1c evaluation

SUMMARY:
This study aims to assess analytical performance of four BGMs and four HbA1c POC devices in comparison to suitable comparator or reference methods, with the view to evaluate performance in the hands of trained users, as well as intended users who are unfamiliar with the system (lay users, for BGMs only). System usability will also be assessed for all BGMs (including lancing devices) and HbA1c devices.

ELIGIBILITY:
Inclusion Criteria:

Arm 1:

* 13-17 years, diagnosed with diabetes and able to manage condition independently (ideally at least 10% of total Arm 1 population)

  •≥18 years, diagnosed with diabetes
* Able and willing to provide informed consent/assent
* Naïve to the SMBG use of the investigational devices
* 10% naïve to any SMBG (defined as not having performed any SMBG in the last 24 months)
* Haematocrit within 20-60%
* Pre-screen BGM result qualifies for inclusion in any of the five glucose concentration ranges based on % of subjects required to meet the target number per concentration range

Arm 2:

•≥18 years

* Able and willing to provide informed consent
* Diagnosed or not diagnosed with diabetes
* Haemoglobin values ≥ 8g/dL
* Pre-screen HbA1c result qualifies for inclusion in the target HbA1c range and % of subjects required for the mid-range values

Exclusion Criteria:

Arm 1:

* <13 years
* 13-17 years and not diagnosed with diabetes or unable to manage condition independently
* Previous use of investigational BGM for SMBG
* Haematocrit outside normal range
* Pre-screen BGM result falling in a glucose concentration range that already has sufficient participants.

Arm 2:

* <18 years
* Haemoglobin value < 8g/dL
* Pre-screen HbA1c result falling in a concentration range that already has sufficient participants.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 910 (Estimated)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
BGM Performace | 1 year
  For BGMs: Performance accuracy is based on ISO 15197 criteria, mean relative bias, 95% limits of agreement, and regression slopes of each BGM with respect to two independently validated comparator BGMs (each investigational BGM will be compared to each comparator BGMs independently).
HbA1c Performance | 1 year
  For HbA1c: Performance accuracy is based on regression slopes, mean relative bias, 95% limits of agreement, and of each HbA1c device versus the reference method and the concordance between capillary and venous blood results.

SECONDARY OUTCOMES:
Comprehension | 1 year
  Proportion of label comprehension, system usability and result/symbol interpretation scale rating per question across all lay users stratified by BGM and lancing device; Total system usability score scale per BGM and lancing device.
Usability | 1 year
  Proportion of system usability and result/symbol interpretation scale rating per question across all lay users stratified by BGM and lancing device; Total system usability score scale per BGM and lancing device.
Interpretation | 1 year
  Proportion of result/symbol interpretation scale rating per question across all lay users stratified by BGM and lancing device; Total system usability score scale per BGM and lancing device
Number of errors as observed | 1 year
  Number and type of errors observed; proportion of error type observed per BGM and lancing device .
Type of errors as observed | 1 year
  Number and type of errors observed; proportion of error type observed per BGM and lancing device .
Proportion of label comprehension | 1 year
  Proportion of system usability scale rating per question across all healthcare professionals, stratified by HbA1c POC device; Total system usability score scale per HbA1c POC device
Number of errors as displayed. | 1 year
  Number and type of errors as displayed on the BGM or HbA1c POC devices, stratified by type of user (BGMs only) and device
Type of errors as displayed | 1 year
  Number and type of errors as displayed on the BGM or HbA1c POC devices, stratified by type of user (BGMs only) and device

CONTACTS AND LOCATIONS:
Overall Officials: Priyanka Singh, Study Director — Foundation for Innovative New Diagnostics (FIND)
Locations (3):
- Sihanouk Hospital Centre of Hope, Phnom Penh, Cambodia
- Asociación Colombiana de Diabetes, Bogotá, Bogota D.C., Colombia
- Lagos University Teaching Hospital, Lagos, Nigeria

IPD SHARING:
Plan to Share IPD: No